CLINICAL TRIAL: NCT05464953
Title: Alazher University Dean
Brief Title: Suprachoroidal Triamcinolone Versus Posterior Subtenon Triamcinolone Alone or Formulated in the Management of Diabetic Macular Edema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSTA and DME
Record Dates: First submitted 2022-07-17; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Macular Edema of Left Eye
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formulated Posterior Sub Tenon Triamcinolone (Active Comparator)
  Interventions: Drug: Formulated Triamcinolone
- Posterior Sub Tenon Triamcinolone alone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide
- suprachoroidal Triamcinolone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide is a corticosteroid that has antiangiogenic and anti-inflammatory effects that can inhibit the expression of VEGF and other proinflammatory cytokines, improving best-corrected visual acuity and decreasing central retinal thickness (CRT) in patients with macular edema
  Arms: Posterior Sub Tenon Triamcinolone alone; suprachoroidal Triamcinolone
Drug: Formulated Triamcinolone — Formulated Triamcinolone: is triamcinolone and sodium hyaluronate and chondroitin sulfate
  Arms: Formulated Posterior Sub Tenon Triamcinolone

SUMMARY:
Background Retinal vascular disorders, such as diabetic retinopathy, hypertensive retinopathy, retinal hemorrhage, and retinal vein occlusion are significant causes of vision impairment and blindness worldwide. Diabetic retinopathy (DR) is the most common retinal vascular disorder and is the leading cause of vision loss among patients aged 25 to 74 years.

Aim to compare formulated Posterior Subtenon Triamcinolone acetonide (PSTA) injection versus Posterior Subtenon Triamcinolone acetonide alone versus suprachoroidal triamcinolone in the management of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diminution of vision due to diabetic macular edema.
* CMT ≥ 250 µ.
* Willing to participate in the study.

Exclusion Criteria:

* Unwilling to participate in the study, 2)
* Ischemic RVO,
* previous laser treatment
* Glaucoma, macular ischemia, cataract, vitreous hemorrhage, and neovascularization of the iris,
* patients with previous anti VEGFs or steroid injections or any eye surgery three months before the inclusion,
* Cardiac co-morbidities result in significant hemodynamic changes, 7)Respiratory diseases need treatment with antibiotics,
* Suffering from other chronic diseases as diabetes,
* Patient with allergy from triamcinolone acetonide.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
BCVA | Base line
  Best-corrected visual acuity
BCVA | at 1st month
  Best-corrected visual acuity
BCVA | at 3rd month
  Best-corrected visual acuity
BCVA | at 6th month
  Best-corrected visual acuity
CMT | at baseline
  CENTRAL MACULAR THICKNESS
CMT | at 1st month
  CENTRAL MACULAR THICKNESS
CMT | at 3rd month
  CENTRAL MACULAR THICKNESS
CMT | at 6th month
  CENTRAL MACULAR THICKNESS

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided